CLINICAL TRIAL: NCT02661204
Title: Diagnostic Performance of an Automated Breast Ultrasound System (ABUS): a Single Centre Study
Brief Title: Diagnostic Performance of an Automated Breast Ultrasound System (ABUS)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: BASEC 2015-00011
Record Dates: First submitted 2016-01-13; First posted 2016-01-22 (Estimated); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer; Implants
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Population A: Consecutive women in the age range 20 to 40 years, with a strong family history of breast cancer or a predisposing gene mutation such as BRCA1 or BRCA2, referring to our department for breast evaluation with ultrasound, will be invited to participate to the study. During the interview, before imaging examination, women will be questioned about family history as well as other relevant personal information (e.g. previous surgery or biopsy for benign breast disease).
  Interventions: Device: Automated breast ultrasound examination (ABUS)
- Population B: Consecutive women with a new breast cancer diagnosis and undergoing pre-operative MRI examination for local staging will be invited to participate to the study. ABUS will be performed within two weeks before the scheduled surgery.
  Interventions: Device: Automated breast ultrasound examination (ABUS)
- Population C: Consecutive women with BI-RADS 3 and 4 lesions detected in a routine breast imaging examination will be invited to participate to the study. ABUS will be performed just after the routine HH-US examination.
  Interventions: Device: Automated breast ultrasound examination (ABUS)
- Population D: Consecutive women undergoing breast MRI examination for the evaluation of breast implants integrity will be invited to participate to the study. ABUS will be performed just after the breast MRI.
  Interventions: Device: Automated breast ultrasound examination (ABUS)

INTERVENTIONS:
Device: Automated breast ultrasound examination (ABUS) — Automated breast ultrasound examination

SUMMARY:
The purpose of this study is to evaluate the diagnostic performance of a new ABUS system among 4 different population:

Population A: women undergoing screening for familial or genetic predisposition for breast cancer.

Population B: women with newly diagnosed breast cancer. ABUS performance will be compared to breast MRI in the pre-operative assessment of breast cancer extent.

Population C: women with BI-RADS 3 or 4 lesions in a routine breast imaging examination. ABUS will be evaluate as a problem-solving tool.

Population D: women undergoing breast MRI for the assessment of breast implants integrity. ABUS performance will be compared to breast MRI.

DETAILED DESCRIPTION:
Population A: women in the age range of 20 to 40 years, with a strong family history of breast cancer or a predisposing gene mutation such as BRCA1 or BRCA2. A total of 100 patients should be enrolled.

Population B: women with new breast cancer diagnosis undergoing pre-operative local cancer staging.A total of 50 patients will be enrolled.

Population C: women with lesions classified BI-RADS 3 or 4 in a routine breast imaging examination. A total of 50 patients will be enrolled.

Population D: women undergoing breast-MRI for the evaluation of breast implants integrity. A total of 50 patients will be enrolled.

The expected duration of subject participation is 5 years for population A: every year the patients will undergo ABUS examination and the results will be compared with HHUS examination.

In population B, C and D only one examination will be performed and the data obtained with ABUS will be compared with HH-US and breast MRI data.

Images will be evaluated by a radiologist with breast imaging experience and ABUS findings will be compared with findings from HHUS and MR imaging.

Afterwards, two or three readers (radiologists with different levels of experience in breast imaging) blinded to clinical, HH-US and MRI data, will evaluate the interobserver agreement ABUS images will be evaluated by Methods of minimising bias Population A - During the recruitment, family history of breast cancer will be in-depth analysed in order to avoid the bias related to different levels of risk for breast cancer. In order to reduce the loss of patients to follow-up, women will be invited every year to undergo HHUS and ABUS examination at our department.

ELIGIBILITY:
Inclusion Criteria:

1. Population A - Inclusion criteria:

   * Age between 20 and 40 years
   * family history of breast cancer or a proved predisposing gene mutation such as BRCA1 or BRCA2
2. Population B - Inclusion criteria

   * Age ≥ 18 years
   * Newly diagnosed breast cancer with no previous history of breast cancer
   * Availability of pre-operative breast MRI performed for local staging within 4 weeks before the surgery
   * Breast surgery performed at the UniversitätsSpital Zürich
3. Population C - Inclusion criteria

   * Age ≥ 18 years
   * Newly detected BI-RADS 3 or 4 lesion
   * Availability of follow-up examination or histological results of biopsy and surgery
4. Population D - Inclusion criteria

   * Age ≥ 18 years
   * Availability of breast MRI performed for evaluating breast implants integrity

Exclusion Criteria:

1) Population A - Exclusion criteria:

* Personal history of breast or ovarian cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population A: women in the age range of 20 to 40 years, with a strong family history of breast cancer or a predisposing gene mutation such as BRCA1 or BRCA2. A total of 100 patients should be enrolled.
  Population B: women with new breast cancer diagnosis undergoing pre-operative local cancer staging.A total of 50 patients will be enrolled.
  Population C: women with lesions classified BI-RADS 3 or 4 in a routine breast imaging examination. A total of 50 patients will be enrolled.
  Population D: women undergoing breast-MRI for the evaluation of breast implants integrity. A total of 50 patients will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2016-01; Primary Completion 2023-05 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Population A: comparison between ABUS and HHUS with respect to the number of lesions detected with the two devices and their characterization according to the BI-RADS lexicon | 5 years
Population B:comparison between ABUS and breast MRI with respect to known malignant lesion/s size assessment and number of additional lesions detected and not previously evident with mammography and HHUS | 5 years
  sensitivity and specificity of a new ABUS system in the assessment of breast cancer extent. Breast MRI will be used as standard of reference
Population C: number of patients with diagnosis of BI-RADS 3 and 4 breast lesions with ABUS compared to histological results or follow-up | 5 years
  sensitivity and specificity of a new ABUS system in the assessment of BI-RADS 3 and 4 lesions. Follow-up and histological results of the biopsy or surgery will be used as standard of reference
Population D: number of participants with suspected rupture of breast implants diagnosed with ABUS compared to breast MRI diagnosis | 5 years
  sensitivity and specificity of a new ABUS system in the assessment of breast implants integrity. Breast MRI will be used as standard of reference

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Boss, MD, Principal Investigator — University Hospital Zurich, Institute of Diagnostic and Interventional Radiology, University Hospital Zurich
Locations (1):
- University Hospital Zurich, Institute of Diagnostic and Interventional Radiology, University Hospital Zurich, Zurich, Switzerland